CLINICAL TRIAL: NCT03711149
Title: Randomized Controlled Trial of Activity Monitor Feedback and Interactive Ambulation Tours to Improve Postoperative Ambulation and Efficiency Outcomes After Major Surgery
Brief Title: Activity Monitor Feedback and Interactive Tours to Improve Postoperative Ambulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Timothy J. Daskivich, Director of Health Services Research, Department of Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00051802
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Surgery
Keywords: Ambulation; Length of stay; Patient Satisfaction; Activity Monitor; Digital Health
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial will involve two arms: (1) and intervention arm consisting of activity monitor feedback loop and art tours and (2) control group consisting of standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention: Activity monitor feedback loop: (1) Subjects will receive activity monitor with feedback on daily step count from the in-room TV screen, and (2) access to the Art Tour application
  Interventions: Other: Activity monitor feedback loop
- Standard-of-care Arm (No Intervention): Subjects in the control arm will receive a "blinded" activity monitor post-op (without feedback on step count) and the usual standard of care. Nurses and doctors will not monitor ambulation with the activity monitor, they will use standard methods of observation.

INTERVENTIONS:
Other: Activity monitor feedback loop — The intervention arm will test if the feedback system (i.e., activity monitor, real-time feedback, and art tours) increases daily step count, decreases length of stay, and improves patient and provider communication, patient awareness of step count goals, and patient confidence in accomplishment of daily goals.
  Arms: Intervention Arm

SUMMARY:
This is a randomized controlled trial that compares a system using activity monitors to provide real-time feedback on daily ambulation to patients undergoing major surgeries, paired with step-count-measured art tours of the surgical units, versus standard of care, on step count. The hypothesis is that the feedback system + art tours will encourage patients to ambulate more.

DETAILED DESCRIPTION:
After major surgery, patients are encouraged to walk early and often, since early ambulation is linked with improved clinical and efficiency outcomes. This research study tests whether providing goal-directed feedback on daily ambulation to patients using activity monitors in combination with an app that provides step count-rated "art tours" of the surgical floors will increase the amount of steps taken after surgery. Upon enrollment, all patients will be assigned to either the control (no intervention) or experimental (activity monitor feedback + art tours) group, stratified by surgery type. This randomized controlled trial aims to determine if this feedback system/art tours approach improves: (1) daily step count, (2) length of stay, and (3) patient satisfaction compared with standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing one of the 14 surgeries: Gynecological (Total Abdominal Hysterectomy, Gyn Ex Lap); Orthopedic (Total Hip Replacement, Total Knee Replacement); Minimally Invasive Surgery (Hiatal Hernia Repair/Fundoplication, Gastric Bypass, Gastric Sleeve); Colorectal Surgery (Lap/Robotic Colectomy, Ileocolic Resection, Open Colectomy); Thoracic (Lung Lobectomy); Urologic (Robotic Cystectomy, Radical Prostatectomy, Partial Nephrectomy).
* Able to provide informed consent
* Non-English speakers will be included with the use of short forms in the 7 available languages
* Must have access to an IOS or Android device

Exclusion Criteria:

* Unable to provide consent
* Not undergoing procedure of interest
* Admitted to ICU directly after operation (except esophagectomy, where all patients are admitted to ICU directly after the operation)
* Use of walker, cane, or wheelchair at baseline
* Presence of physical limitations on walking (i.e. amputation)
* Usual place of residence is skilled nursing facility
* Cognitive inability to follow directions to maintain activity monitor in place
* Unable to place activity monitor on patient's wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-10-22 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Daily Step Count | During hospitalization within approximately 1-2 weeks
  Daily step count will be captured with activity monitor

SECONDARY OUTCOMES:
Length of stay | Within approximately 1-2 weeks, Date patient was admitted through hospital discharge
  Length of stay in intervention arm compared to control
Patient Satisfaction | Within approximately 1-2 weeks, Day patient is discharged from hospital
  Patient satisfaction measured using likert-scale rated items. Scale measures patient/physician communication, patient awareness of step goals, and patient confidence in accomplishment of daily goals. The following scale ranges will be used:
  1. Never, Once a day, Twice a day, Three times a day, More than three times a day
  2. Much lower, Lower, About the same, Higher, Much higher
  3. Not at all, Slightly, Moderately, Very, Extremely
  Positive answer in likert-scales indicate higher patient/physician communication, patient awareness, and patient confidence in accomplishing daily step goals.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Daskivich, MD, MSHPM, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States